CLINICAL TRIAL: NCT04925232
Title: Transcranial Magnetic Stimulation for Visual Snow Syndrome: An Open-Label Feasibility Treatment Trial
Brief Title: Transcranial Magnetic Stimulation For Visual Snow Syndrome
Acronym: TMSVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-0424
Record Dates: First submitted 2021-05-17; First posted 2021-06-14 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Visual Snow Syndrome
Keywords: repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — visual snow syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- One group (Experimental): All participants will undergo 2 weeks (5 times each week) of repetitive TMS
  Interventions: Device: Transcranial Magnetic Stimulation device

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation device — Five days a week for 2 consecutive weeks, participants will have repetitive TMS at specific paramaters
  Other Names: TMS

SUMMARY:
This study aims to investigate the feasibility of the use of repetitive transcranial magnetic stimulation (rTMS) for symptoms associated with Visual Snow syndrome (VS).

DETAILED DESCRIPTION:
The study will gather information about the treatment of up to 10 people with VS using rTMS. Treated participants will undergo 10 sessions of rTMS administered 5 times a week over 2 weeks. All visits will take place in the University of Colorado School of Medicine NeuroMag/Transcranial Magnetic Stimulation laboratory on University of Colorado Anschutz Medical Campus.

The specific aims for this feasibility study include:

1. Determine whether any participant experiences untoward effects of rTMS in the setting of visual snow syndrome and determine the potential drop-out rate of larger study.
2. Determine the performance of a novel scale (Colorado Visual Snow Scale) and two three psychophysical visual processing tasks

   1. Determine the standard deviation and test-retest reliability for the novel scale and two visual processing tasks
   2. Determine whether the visual processing tasks perform similar to performance found by the developer
3. Describe changes in outcome measures between pre- and post-treatment with rTMS

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of VS that meets International Headache Society criteria
* Able to provide meaningful informed consent
* Visual snow must be present for more than three months and must be persistent (i.e. continuous)
* A prior clinical Brain MRI with and without contrast done in the past 3 years that does not show signs of clinically significant brain lesions (no evidence of multiple sclerosis, stroke, brain tumor, cortical heterotopia or other cortical developmental abnormalities, arteriovenous malformation, etc…)

Exclusion Criteria:

* Syndrome meeting criteria for Hallucinogen-persisting perception disorder
* Prior treatment with TMS for any disorder
* Epilepsy, family history of epilepsy, or personal history of seizure
* Any medical condition or medication that increases the risk of seizure
* Pacemaker or other implantable medical device
* Metal in the skull, not including the mouth
* Unstable cardiac, pulmonary, or other systemic illness
* Pregnancy
* Bipolar disorder
* History of suicidality

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
TMS Side Effect Questionnaire | Week 1
  The TMS Side Effect Questionnaire queries participants for specific and potential side effects related to TMS. It also allows for open ended answers regarding potential side effects from TMS. The percent of participants experiencing adverse events directly related to treatment will be reported.
TMS Side Effect Questionnaire | Week 2
  The TMS Side Effect Questionnaire queries participants for specific and potential side effects related to TMS. It also allows for open ended answers regarding potential side effects from TMS.The percent of participants experiencing adverse events directly related to treatment will be reported.
TMS Side Effect Questionnaire | Month 1
  The TMS Side Effect Questionnaire queries participants for specific and potential side effects related to TMS. It also allows for open ended answers regarding potential side effects from TMS.The percent of participants experiencing adverse events directly related to treatment will be reported.
TMS Side Effect Questionnaire | Month 3
  The TMS Side Effect Questionnaire queries participants for specific and potential side effects related to TMS. It also allows for open ended answers regarding potential side effects from TMS. The percent of participants experiencing adverse events directly related to treatment will be reported.
Visual Noise Task | Week 1
  This task will assess physiological properties of the visual system related to visual noise and will measure luminance increment detection threshold in a noise task with scores from 0-7, with higher scores considered poorer performance.
Visual Noise Task | Week 2
  This task will assess physiological properties of the visual system related to visual noise and will measure luminance increment detection threshold in a noise task with scores from 0-7, with higher scores considered poorer performance.
Visual Noise Task | Month 1
  This task will assess physiological properties of the visual system related to visual noise and will measure luminance increment detection threshold in a noise task with scores from 0-7, with higher scores considered poorer performance.
Visual Noise Task | Month 3
  This task will assess physiological properties of the visual system related to visual noise and will measure luminance increment detection threshold in a noise task with scores from 0-7, with higher scores considered poorer performance.
Visual Contrast Task | Week 1
  This task will assess physiological properties of the visual system related to contrast and will measure the suppression index for a center-surround suppression task with scores from -1.00 to +1.00, with lower scores considered poorer performance
Visual Contrast Task | Week 2
  This task will assess physiological properties of the visual system related to contrast and will measure the suppression index for a center-surround suppression task with scores from -1.00 to +1.00, with lower scores considered poorer performance
Visual Contrast Task | Month 1
  This task will assess physiological properties of the visual system related to contrast and will measure the suppression index for a center-surround suppression task with scores from -1.00 to +1.00, with lower scores considered poorer performance
Visual Contrast Task | Month 3
  This task will assess physiological properties of the visual system related to contrast and will measure the suppression index for a center-surround suppression task with scores from -1.00 to +1.00, with lower scores considered poorer performance
Global Motion Task | Week 1
  Each test will assess physiological properties of the visual system related to global motion and measure pattern coherence threshold for global motion task with scores from 0.00 to 1.00, with higher thresholds considered poorer performance.
Global Motion Task | Week 2
  Each test will assess physiological properties of the visual system related to global motion and measure pattern coherence threshold for global motion task with scores from 0.00 to 1.00, with higher thresholds considered poorer performance.
Global Motion Task | Month 1
  Each test will assess physiological properties of the visual system related to global motion and measure pattern coherence threshold for global motion task with scores from 0.00 to 1.00, with higher thresholds considered poorer performance.
Global Motion Task | Month 3
  Each test will assess physiological properties of the visual system related to global motion and measure pattern coherence threshold for global motion task with scores from 0.00 to 1.00, with higher thresholds considered poorer performance.
Colorado Visual Snow Symptom Scale | Week 1
  Colorado Visual Snow Scale is a novel scale created for this study and to investigate its use in measure symptom severity. There are 11 subscales: Visual Static, Afterimages, Trails, Blue Field Entoptic Phenomenon, Floaters, Night Vision Problems, Tinnitus, Feeling of Detachment, Anxiety, Depression, Sleep Issues. Each section assess symptom severe, impact on vision, impact on daily activities, and ability to drive with scale of 0-10 wiht 10 being more severe or impairing the symptom. Total score for each subscale can range from 0-40 and total score overall can range from 0-440 and the higher the score the more severe or impairing the symptoms.
Colorado Visual Snow Symptom Scale | Week 2
  Colorado Visual Snow Scale is a novel scale created for this study and to investigate its use in measure symptom severity. There are 11 subscales: Visual Static, Afterimages, Trails, Blue Field Entoptic Phenomenon, Floaters, Night Vision Problems, Tinnitus, Feeling of Detachment, Anxiety, Depression, Sleep Issues. Each section assess symptom severe, impact on vision, impact on daily activities, and ability to drive with scale of 0-10 wiht 10 being more severe or impairing the symptom. Total score for each subscale can range from 0-40 and total score overall can range from 0-440 and the higher the score the more severe or impairing the symptoms.
Colorado Visual Snow Symptom Scale | Month 1
  Colorado Visual Snow Scale is a novel scale created for this study and to investigate its use in measure symptom severity. There are 11 subscales: Visual Static, Afterimages, Trails, Blue Field Entoptic Phenomenon, Floaters, Night Vision Problems, Tinnitus, Feeling of Detachment, Anxiety, Depression, Sleep Issues. Each section assess symptom severe, impact on vision, impact on daily activities, and ability to drive with scale of 0-10 wiht 10 being more severe or impairing the symptom. Total score for each subscale can range from 0-40 and total score overall can range from 0-440 and the higher the score the more severe or impairing the symptoms.
Colorado Visual Snow Symptom Scale | Month 3
  Colorado Visual Snow Scale is a novel scale created for this study and to investigate its use in measure symptom severity. There are 11 subscales: Visual Static, Afterimages, Trails, Blue Field Entoptic Phenomenon, Floaters, Night Vision Problems, Tinnitus, Feeling of Detachment, Anxiety, Depression, Sleep Issues. Each section assess symptom severe, impact on vision, impact on daily activities, and ability to drive with scale of 0-10 wiht 10 being more severe or impairing the symptom. Total score for each subscale can range from 0-40 and total score overall can range from 0-440 and the higher the score the more severe or impairing the symptoms.
Drop out rate | Month 3
  The number of participants who drop out will be determined at the end of the study.
Visual Functional Quality Scale (VFQ-25) | Week 1
  The VFQ-25 is a reliable and valid 25-item version of the 51-item National Eye Institute Visual Function Questionnaire (NEI-VFQ) and it is useful in clinical trials to measure quality of visual functioning. Scores range from 0-100 with higher scores indicating better quality visual functioning in everyday activities.
Visual Functional Quality Scale (VFQ-25) | Week 2
  The VFQ-25 is a reliable and valid 25-item version of the 51-item National Eye Institute Visual Function Questionnaire (NEI-VFQ) and it is useful in clinical trials to measure quality of visual functioning. Scores range from 0-100 with higher scores indicating better quality visual functioning in everyday activities.
Visual Functional Quality Scale (VFQ-25) | Month 1
  The VFQ-25 is a reliable and valid 25-item version of the 51-item National Eye Institute Visual Function Questionnaire (NEI-VFQ) and it is useful in clinical trials to measure quality of visual functioning. Scores range from 0-100 with higher scores indicating better quality visual functioning in everyday activities.
Visual Functional Quality Scale (VFQ-25) | Month 3
  The VFQ-25 is a reliable and valid 25-item version of the 51-item National Eye Institute Visual Function Questionnaire (NEI-VFQ) and it is useful in clinical trials to measure quality of visual functioning. Scores range from 0-100 with higher scores indicating better quality visual functioning in everyday activities.
General Anxiety Disorder Scale (GAD-7) | Week 1
  Screening questionnaire that measures the degree of anxiety with scores ranging from 0-21 and higher scores indicate greater anxiety. Scores of 5, 10, and 15 can be interpreted as representing mild, moderate, and severe levels of anxiety.
General Anxiety Disorder Scale (GAD-7) | Week 2
  Screening questionnaire that measures the degree of anxiety with scores ranging from 0-21 and higher scores indicate greater anxiety. Scores of 5, 10, and 15 can be interpreted as representing mild, moderate, and severe levels of anxiety.
General Anxiety Disorder Scale (GAD-7) | Month 1
  Screening questionnaire that measures the degree of anxiety with scores ranging from 0-21 and higher scores indicate greater anxiety. Scores of 5, 10, and 15 can be interpreted as representing mild, moderate, and severe levels of anxiety.
General Anxiety Disorder Scale (GAD-7) | Month 3
  Screening questionnaire that measures the degree of anxiety with scores ranging from 0-21 and higher scores indicate greater anxiety. Scores of 5, 10, and 15 can be interpreted as representing mild, moderate, and severe levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — CU School of Medicine
Locations (1):
- University of Colorado School of Medicine Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Protocol will be published

REFERENCES:
- [Derived] Grande M, Lattanzio L, Buard I, McKendrick AM, Chan YM, Pelak VS. A Study Protocol for an Open-Label Feasibility Treatment Trial of Visual Snow Syndrome With Transcranial Magnetic Stimulation. Front Neurol. 2021 Sep 24;12:724081. doi: 10.3389/fneur.2021.724081. eCollection 2021. PMID 34630299